CLINICAL TRIAL: NCT05726695
Title: The Use of miRNA Detection for Diagnostics of Cardiovascular Diseases
Brief Title: The Use of Blood Biochemical Markers for Diagnostics of Heart Muscle Diseases
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: miRNA-RVO-FNOs/2018-05KVO; RVO-FNOs/2018-05KVO (Other Grant/Funding Number: University Hospital Ostrava)
Record Dates: First submitted 2019-08-01; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure; Heart Dilation; Left Ventricular Hypertrophy
Keywords: microRNA; immunomethods; heart failure biomarkers
MeSH Terms: conditions — Heart Failure; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Full blood samples, no DNA examination will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heart failure with reduced ejection fraction.: Patients indicated for biochemical analysis due to a suspected heart disease, with HFrEF diagnosed on echocardiography with left-ventricular ejection fraction lower than 35%.
  Diagnostic Test: MicroRNA test. Laboratory analysis for the detection of microRNA in blood samples.
  Diagnostic Test: Heart ultrasound examination. Heart ultrasound examination will be performed as a standard cardiology examination.
  Interventions: Diagnostic Test: microRNA test; Diagnostic Test: Heart ultrasound examination
- Control group: Patients with no known heart disease (hypertrophy or dilatation), which has been confirmed on echocardiography.
  Diagnostic Test: microRNA test. Laboratory analysis for the detection of microRNA in blood samples.
  Diagnostic Test: Heart ultrasound examination. Heart ultrasound examination will be performed as a standard cardiology examination.
  Interventions: Diagnostic Test: microRNA test; Diagnostic Test: Heart ultrasound examination

INTERVENTIONS:
Diagnostic Test: microRNA test — Laboratory analysis for the detection of microRNA in blood samples.
Diagnostic Test: Heart ultrasound examination — Heart ultrasound examination will be performed as a standard cardiology examination.

SUMMARY:
The aim of the study is to determine the analytical characteristics of the microRNA enzymatic immunoassay (miREIA) method and to determine various relations among miRNA biomarkers and heart failure (HF) with reduced ejection fraction(HFrEF).

The investigators assume that there are correlations between levels of selected miRNA and HFrEF. These correlations provide information to formulate pathophysiological conclusions, which will significantly contribute to early diagnostics and also the treatment of this disease.

DETAILED DESCRIPTION:
Heart failure presents a significant diagnostic and treatment problem. The mortality in the Czech Republic related to this condition is high. The current treatment strategy consists of the administration of medication to patients, in order to attenuate the clinical manifestations of the disease and to influence the overall survival of patients suffering from this condition. Another treatment option is a mini-invasive procedure, with implantation of a pacemaker with biventricular stimulation, or transplantation of the heart. Despite these treatment options, the mortality of patients due to heart failure remains high, and new approaches are being studied for the diagnostics and treatment of heart failure. Factors that may play an important role in earlier diagnostics are miRNA. These molecules are located in the circulating blood. They are being described as suitable prognostic markers of heart failure, which may contribute to earlier diagnostics and bring a better understanding of processes going on in the human body.

In the study, the authors will take blood samples in order to analyze the presence of miRNA. These levels of miRNA will be compared with heart ultrasound parameters of HF patients and healthy control subjects.

ELIGIBILITY:
Inclusion criteria (patient group):

* left ventricle ejection fraction (EF LV) equal or less than 40%
* age between 18-80 years

Inclusion criteria (control group):

* normal EF LV (left ventricular ejection fraction)
* no structural cardiac abnormalities
* age between 18-80 years.

Exclusion criteria:

* recent myocardial infarction
* recent percutaneous coronary intervention (PCI)
* recent decompensation of chronic heart failure
* chronic kidney disease with need for haemodialysis
* creatin level over 450 umol/l
* signs of acute or chronic inflammation with CRP (C-reactive protein) over 20 mg/l
* patient with a known tumour
* history of cardiovascular disease
* diabetes mellitus
* severe liver and kidney disease
* BNP (brain natriuretic peptide) > 250 pg/ml or NTproBNP > 500 pg/ml for males and 750 pg/ml for females
* signs of acute or chronic inflammation with CRP over 20 mg/l

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known stable heart failure hospitalized or followed at the outpatient clinic at the University Hospital Ostrava, Department of Cardiovascular Diseases.
  The control group consists of healthy individuals, who had volunteered for the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Levels of miRNA (in pmol/L) | 43 months
  Full blood samples will be taken in both groups after period of clinically stable state and analyzed for levels of miRNA(hsa-miR-21-5p; hsa-miR-23a-3p; hsa-miR-142-5p; hsa-miR-126-3p) with biochemical microRNA enzymatic immunoassay. Measured levels of listed four miRNAs will be provided pmol/L.
  These levels will be statistically analyzed and compared between patient and control group.

SECONDARY OUTCOMES:
Correlation between miRNA levels and 1-year mortality and risk of rehospitalization | 43 months
  We will examine levels of miRNA in corelation to 1-year mortality and risk of rehospitalization acquired from Czech national registry (UZIS).

CONTACTS AND LOCATIONS:
Overall Officials: Lukáš Evin, MD,Ph.D., Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava-Poruba, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Catalanotto C, Cogoni C, Zardo G. MicroRNA in Control of Gene Expression: An Overview of Nuclear Functions. Int J Mol Sci. 2016 Oct 13;17(10):1712. doi: 10.3390/ijms17101712. PMID 27754357
- [Background] Bartel DP. MicroRNAs: genomics, biogenesis, mechanism, and function. Cell. 2004 Jan 23;116(2):281-97. doi: 10.1016/s0092-8674(04)00045-5. PMID 14744438
- [Background] Lim LP, Lau NC, Garrett-Engele P, Grimson A, Schelter JM, Castle J, Bartel DP, Linsley PS, Johnson JM. Microarray analysis shows that some microRNAs downregulate large numbers of target mRNAs. Nature. 2005 Feb 17;433(7027):769-73. doi: 10.1038/nature03315. Epub 2005 Jan 30. PMID 15685193
- [Background] Chen X, Ba Y, Ma L, Cai X, Yin Y, Wang K, Guo J, Zhang Y, Chen J, Guo X, Li Q, Li X, Wang W, Zhang Y, Wang J, Jiang X, Xiang Y, Xu C, Zheng P, Zhang J, Li R, Zhang H, Shang X, Gong T, Ning G, Wang J, Zen K, Zhang J, Zhang CY. Characterization of microRNAs in serum: a novel class of biomarkers for diagnosis of cancer and other diseases. Cell Res. 2008 Oct;18(10):997-1006. doi: 10.1038/cr.2008.282. PMID 18766170
- [Background] Weber JA, Baxter DH, Zhang S, Huang DY, Huang KH, Lee MJ, Galas DJ, Wang K. The microRNA spectrum in 12 body fluids. Clin Chem. 2010 Nov;56(11):1733-41. doi: 10.1373/clinchem.2010.147405. Epub 2010 Sep 16. PMID 20847327
- [Background] Turchinovich A, Weiz L, Langheinz A, Burwinkel B. Characterization of extracellular circulating microRNA. Nucleic Acids Res. 2011 Sep 1;39(16):7223-33. doi: 10.1093/nar/gkr254. Epub 2011 May 24. PMID 21609964
- [Background] Zernecke A, Bidzhekov K, Noels H, Shagdarsuren E, Gan L, Denecke B, Hristov M, Koppel T, Jahantigh MN, Lutgens E, Wang S, Olson EN, Schober A, Weber C. Delivery of microRNA-126 by apoptotic bodies induces CXCL12-dependent vascular protection. Sci Signal. 2009 Dec 8;2(100):ra81. doi: 10.1126/scisignal.2000610. PMID 19996457
- [Background] Tabet F, Vickers KC, Cuesta Torres LF, Wiese CB, Shoucri BM, Lambert G, Catherinet C, Prado-Lourenco L, Levin MG, Thacker S, Sethupathy P, Barter PJ, Remaley AT, Rye KA. HDL-transferred microRNA-223 regulates ICAM-1 expression in endothelial cells. Nat Commun. 2014 Feb 28;5:3292. doi: 10.1038/ncomms4292. PMID 24576947
- [Background] Vickers KC, Palmisano BT, Shoucri BM, Shamburek RD, Remaley AT. MicroRNAs are transported in plasma and delivered to recipient cells by high-density lipoproteins. Nat Cell Biol. 2011 Apr;13(4):423-33. doi: 10.1038/ncb2210. Epub 2011 Mar 20. PMID 21423178
- [Background] Arroyo JD, Chevillet JR, Kroh EM, Ruf IK, Pritchard CC, Gibson DF, Mitchell PS, Bennett CF, Pogosova-Agadjanyan EL, Stirewalt DL, Tait JF, Tewari M. Argonaute2 complexes carry a population of circulating microRNAs independent of vesicles in human plasma. Proc Natl Acad Sci U S A. 2011 Mar 22;108(12):5003-8. doi: 10.1073/pnas.1019055108. Epub 2011 Mar 7. PMID 21383194
- [Background] Wang K, Zhang S, Weber J, Baxter D, Galas DJ. Export of microRNAs and microRNA-protective protein by mammalian cells. Nucleic Acids Res. 2010 Nov;38(20):7248-59. doi: 10.1093/nar/gkq601. Epub 2010 Jul 7. PMID 20615901
- [Background] Kosaka N, Iguchi H, Yoshioka Y, Takeshita F, Matsuki Y, Ochiya T. Secretory mechanisms and intercellular transfer of microRNAs in living cells. J Biol Chem. 2010 Jun 4;285(23):17442-52. doi: 10.1074/jbc.M110.107821. Epub 2010 Mar 30. PMID 20353945
- [Background] Zhu H, Fan GC. Extracellular/circulating microRNAs and their potential role in cardiovascular disease. Am J Cardiovasc Dis. 2011 Jul 30;1(2):138-149. PMID 22059153
- [Background] Navickas R, Gal D, Laucevicius A, Taparauskaite A, Zdanyte M, Holvoet P. Identifying circulating microRNAs as biomarkers of cardiovascular disease: a systematic review. Cardiovasc Res. 2016 Sep;111(4):322-37. doi: 10.1093/cvr/cvw174. Epub 2016 Jun 29. PMID 27357636
- [Background] Heggermont WA, Heymans S. MicroRNAs are involved in end-organ damage during hypertension. Hypertension. 2012 Nov;60(5):1088-93. doi: 10.1161/HYPERTENSIONAHA.111.187104. Epub 2012 Sep 17. PMID 22987922
- [Background] Ackerman MJ, Priori SG, Willems S, Berul C, Brugada R, Calkins H, Camm AJ, Ellinor PT, Gollob M, Hamilton R, Hershberger RE, Judge DP, Le Marec H, McKenna WJ, Schulze-Bahr E, Semsarian C, Towbin JA, Watkins H, Wilde A, Wolpert C, Zipes DP. HRS/EHRA expert consensus statement on the state of genetic testing for the channelopathies and cardiomyopathies this document was developed as a partnership between the Heart Rhythm Society (HRS) and the European Heart Rhythm Association (EHRA). Heart Rhythm. 2011 Aug;8(8):1308-39. doi: 10.1016/j.hrthm.2011.05.020. No abstract available. PMID 21787999
- [Background] Jiao M, You HZ, Yang XY, Yuan H, Li YL, Liu WX, Jin M, Du J. Circulating microRNA signature for the diagnosis of childhood dilated cardiomyopathy. Sci Rep. 2018 Jan 15;8(1):724. doi: 10.1038/s41598-017-19138-4. PMID 29335596
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Joladarashi D, Thandavarayan RA, Babu SS, Krishnamurthy P. Small engine, big power: microRNAs as regulators of cardiac diseases and regeneration. Int J Mol Sci. 2014 Sep 9;15(9):15891-911. doi: 10.3390/ijms150915891. PMID 25207600
- [Background] Zhang Y, Liu YJ, Liu T, Zhang H, Yang SJ. Plasma microRNA-21 is a potential diagnostic biomarker of acute myocardial infarction. Eur Rev Med Pharmacol Sci. 2016;20(2):323-9. PMID 26875904
- [Background] Thum T, Gross C, Fiedler J, Fischer T, Kissler S, Bussen M, Galuppo P, Just S, Rottbauer W, Frantz S, Castoldi M, Soutschek J, Koteliansky V, Rosenwald A, Basson MA, Licht JD, Pena JT, Rouhanifard SH, Muckenthaler MU, Tuschl T, Martin GR, Bauersachs J, Engelhardt S. MicroRNA-21 contributes to myocardial disease by stimulating MAP kinase signalling in fibroblasts. Nature. 2008 Dec 18;456(7224):980-4. doi: 10.1038/nature07511. Epub 2008 Nov 30. PMID 19043405
- [Background] Bang C, Batkai S, Dangwal S, Gupta SK, Foinquinos A, Holzmann A, Just A, Remke J, Zimmer K, Zeug A, Ponimaskin E, Schmiedl A, Yin X, Mayr M, Halder R, Fischer A, Engelhardt S, Wei Y, Schober A, Fiedler J, Thum T. Cardiac fibroblast-derived microRNA passenger strand-enriched exosomes mediate cardiomyocyte hypertrophy. J Clin Invest. 2014 May;124(5):2136-46. doi: 10.1172/JCI70577. Epub 2014 Apr 17. PMID 24743145